CLINICAL TRIAL: NCT02060864
Title: Effect of the Enzyme AN-PEP on Gluten Degradation in the Stomach of Gluten-sensitive Individuals
Brief Title: Effect of AN-PEP Enzyme on Gluten Digestion in Gluten Sensitive Individuals
Acronym: AN-PEP-03
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: DSM Food Specialties (Industry)
Responsible Party: Principal Investigator, Robert Brummer, Prof, Örebro University, Sweden
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: AN-PEP-03
Record Dates: First submitted 2014-02-11; First posted 2014-02-12 (Estimated); Last update posted 2015-08-28 (Estimated); Status verified 2015-08

CONDITIONS: Non-coeliac Gluten Sensitivity
Keywords: enzyme; gluten; food intolerance
MeSH Terms: conditions — Food Intolerance

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): 2 Placebo pills
  Interventions: Dietary Supplement: Placebo
- AN-PEP 80.000 PPI (Experimental): 1 pill AN-PEP 80.000 PPI and 1 pill Placebo.
  Interventions: Dietary Supplement: AN-PEP
- AN-PEP 160.000 PPI (Experimental): 2 pills AN-PEP 80.000 PPI
  Interventions: Dietary Supplement: AN-PEP

INTERVENTIONS:
Dietary Supplement: AN-PEP — Two pills are consumed in the morning with a breakfast
  Other Names: Aspergillus Niger-Prolyl Endopeptidase
  Arms: AN-PEP 160.000 PPI; AN-PEP 80.000 PPI
Dietary Supplement: Placebo
  Arms: Placebo

SUMMARY:
In this trial, the effect of a low and a high dose AN-PEP will be investigated in gluten sensitive individuals. Volunteers receive a breakfast with background (0.5 g) gluten. Capsules are taken in the morning within 5 min after start of breakfast. Gastrointestinal fluid will be sampled over 3 hours to measure gluten degradation. After 5 volunteers have completed 3 test days, a blind interim analysis is performed by a third party based on which it is decided whether to proceed with the low AN-PEP dose.

ELIGIBILITY:
Inclusion Criteria:

* Male/female
* Age ≥18 but <70 yr
* Females: Hormonal contraceptive treatment
* Self-reported gluten-sensitive individuals fulfilling the Rome III criteria while consuming gluten
* Subject has read and understood the information provided on the study and given written informed consent

Exclusion Criteria:

* Coeliac disease serology while consuming gluten (serological test for tissue transglutaminase IgA antibodies and total IgA antibodies)
* Wheat allergy (serological test for wheat protein IgE antibodies)
* Medication or medical condition that affects gastric emptying or secretion
* Females: Pregnancy or breast-feeding
* Inability to swallow the gastroduodenal feeding tube
* Any medical condition that in the opinion of the investigators may interfere with the study and may jeopardise the health status of the participant
* Any condition that in the opinion of the investigators may interfere with the study and may jeopardise the health status of the participant

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-04; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Effect of 160.000 PPI AN-PEP on duodenal gluten | 3-hour
  Effect of AN-PEP (160.000 PPI) on gluten degradation based on amount of gluten detected in the duodenum compared with placebo over 180 min (Success is defined as at least 50% gluten degradation compared to placebo in an individual test, calculated using AUC)

SECONDARY OUTCOMES:
Effect of 160.000 PPI AN-PEP on gastric gluten | 3-hour
  Effect of AN-PEP (160.000 PPI) on gluten degradation based on amount of gluten detected in the stomach compared with placebo over 180 min (Success is defined as at least 50% gluten degradation compared to placebo in an individual test, calculated using AUC)
Effect of 80.000 PPI AN-PEP on duodenal gluten | 3-hour
  Effect of AN-PEP (80.000 PPI) on gluten degradation based on amount of gluten detected in the duodenum compared to placebo over 180 min (Success is defined as at least 50% gluten degradation compared to placebo in an individual test, calculated using AUC)
Effect of 80.000 PPI AN-PEP on gastric gluten AUC | 3-hour
  Effect of AN-PEP (80.000 PPI) on gluten degradation based on amount of gluten detected in the stomach compared to placebo over 180 min (Success is defined as at least 50% gluten degradation compared to placebo in an individual test, calculated using AUC)
Effect of 160.000 PPI AN-PEP on percentage duodenal gluten reduction | 3-hour
  The average reduction in gluten concentration (as a continuous measure) following administration of AN-PEP (160.000 PPI) on gluten degradation (defined as the percentage of gluten degraded by 180 minutes) based on gluten detection in the duodenum compared with placebo over 180 min using AUC.
Effect of 160.000 PPI AN-PEP on percentage gastric gluten reduction | 3-hour
  The average reduction in gluten concentration (as a continuous measure) following administration of AN-PEP (160.000 PPI) on gluten degradation (defined as the percentage of gluten degraded by 180 minutes) based on gluten detection in the stomach compared with placebo over 180 min using AUC.
Effect of 80.000 PPI AN-PEP on percentage duodenal gluten reduction | 3-hour
  The average reduction in gluten concentration (as a continuous measure) following administration of AN-PEP (80.000 PPI) on gluten degradation (defined as the percentage of gluten degraded by 180 minutes) based on gluten detection in the duodenum compared with placebo over 180 min using AUC.
Effect of 80.000 PPI AN-PEP on percentage gastric gluten reduction | 3-hour
  The average reduction in gluten concentration (as a continuous measure) following administration of AN-PEP (low and high dose) on gluten degradation (defined as the percentage of gluten degraded by 180 minutes) based on gluten detection in the stomach compared with placebo over 180 min using AUC.

CONTACTS AND LOCATIONS:
Locations (1):
- Örebro University, Örebro, Sweden